CLINICAL TRIAL: NCT01517295
Title: Evaluating the Pharmacokinetic Profile of Hydromorphone in Chronic Pain Patients Taking Hydrocodone/APAP
Brief Title: Pharmacokinetic Study of Hydrocodone/APAP in Chronic Pain Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: NEMA Research, Inc. (Industry)
Collaborators: Medtronic - MITG (Industry); International Clinical Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: NEMA-HydrocodonePK-001
Record Dates: First submitted 2012-01-04; First posted 2012-01-25 (Estimated); Results first posted 2016-07-28 (Estimated); Last update posted 2016-07-28 (Estimated); Status verified 2016-06

CONDITIONS: Chronic Pain
Keywords: Pharmacokinetics; Hydromorphone; Hydrocodone; APAP
MeSH Terms: conditions — Chronic Pain | interventions — Hydrocodone; acetaminophen, hydrocodone drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1 (Experimental): Blood will be drawn at 0, 1, 3, and 5 hours after taking one dose of hydrocodone/APAP. Urine will be taken at hour 0 and 3.
  Interventions: Drug: Hydrocodone
- Group 2 (Experimental): Blood will be drawn at 0, 2, 4, and 6 hours after one dose of hydrocodone/APAP. Urine will be taken at hour 0 and 4.
  Interventions: Drug: Hydrocodone

INTERVENTIONS:
Drug: Hydrocodone — Dose: Standard prescribed dose Frequency: Once Duration: Once
  Other Names: Hydrocodone/APAP; Vicodin

SUMMARY:
Objective is to evaluate the pharmacokinetics profile of hydrocodone's metabolite hydromorphone in patients who are taking hydrocodone on a routine basis for more than 3 months for chronic pain and correlate hydromorphone levels to their hydrocodone usage.

DETAILED DESCRIPTION:
Hydrocodone combinations are the most commonly prescribed pain medications in the United States. All the current available Hydrocodone formulations are short acting and have Acetaminophen/Ibuprofen in them. Chronic pain patients who take pain medications for extended time are overloaded with Acetaminophen and there is a very serious concern about liver failure from excessive concurrent alcohol use. Also all the current hydrocodone combinations available in the U.S. are short acting and provide pain relief for 3-6 hrs.

Hydromorphone is a metabolite of Hydrocodone and plays a significant role in providing pain relief in these patients. Although there are no long acting or extended release hydrocodone formulations that are FDA approve at this time, there is once a day extended release Hydromorphone (ER) approved by FDA and is currently marketed under the name Exalgo ®. PK study of chronic hydrocodone/acetaminophen usage is important to determine equivalent potency with hydromorphone ER, so that clinicians can use a simple conversion formula to switch to hydromorphone ER.

Although medical professionals use the Opiate conversion formula on a regular basis for Opioid rotation, there are no published studies showing the pharmacokinetic data in patients taking hydrocodone for chronic pain.

Our goal is to use this PK data to guide clinicians with this data in using extended release hydromorphone for chronic pain management to provide predictable pain relief and minimize the acetaminophen usage.

ELIGIBILITY:
Inclusion Criteria:

* Man or woman aged 18-75
* Documented clinical diagnosis of chronic pain.
* Have been taking hydrocodone/APAP for their chronic non-cancer pain.
* Subjects currently on hydrocodone/APAP must be taking minimal daily dose of 15mg of Hydrocodone for at least 30 days.
* Subjects must have signed an informed consent document indicating that they understand the purpose of and procedures required for the study and are willing to participate in the study.

Exclusion Criteria:

* Subjects who are taking concomitant medications or Nutraceuticals that interfere with Hydrocodone metabolism as listed in Appendix 11 and/or as deemed clinically significant by a pharmacovigilance team that is contracted to monitor and advise.
* Health concerns that the study physician feels may confound study results.
* Individuals who are cognitively impaired or who are not able to give informed consent.
* Previous participation in a clinical research trial within 30 days prior to randomization.
* The subject has an ongoing abuse of illicit substances, alcohol, or actively smoking marijuana.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2012-02; Primary Completion 2012-05 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Srinivas Nalamachu, MD, Principal Investigator — International Clinical Research Institute; Joseph Pergolizzi, MD, Study Director — NEMA Research, Inc.
Locations (2):
- United States (2):
  - NEMA Research Inc. (CRO), Naples, Florida
  - International Clinical Research Institute, Leawood, Kansas

REFERENCES:
- [Background] Wu Y. [Studies on the analysis of hydrocodone and its metabolite in human urine by GC/MS]. Yao Xue Xue Bao. 1997 Apr;32(4):305-9. Chinese. PMID 11499035
- [Background] Chen YL, Hanson GD, Jiang X, Naidong W. Simultaneous determination of hydrocodone and hydromorphone in human plasma by liquid chromatography with tandem mass spectrometric detection. J Chromatogr B Analyt Technol Biomed Life Sci. 2002 Mar 25;769(1):55-64. doi: 10.1016/s1570-0232(01)00616-x. PMID 11936695
- [Background] Menelaou A, Hutchinson MR, Quinn I, Christensen A, Somogyi AA. Quantification of the O- and N-demethylated metabolites of hydrocodone and oxycodone in human liver microsomes using liquid chromatography with ultraviolet absorbance detection. J Chromatogr B Analyt Technol Biomed Life Sci. 2003 Feb 25;785(1):81-8. doi: 10.1016/s1570-0232(02)00856-5. PMID 12535841
- [Background] Hutchinson MR, Menelaou A, Foster DJ, Coller JK, Somogyi AA. CYP2D6 and CYP3A4 involvement in the primary oxidative metabolism of hydrocodone by human liver microsomes. Br J Clin Pharmacol. 2004 Mar;57(3):287-97. doi: 10.1046/j.1365-2125.2003.02002.x. PMID 14998425
- [Background] Cone EJ, Darwin WD, Gorodetzky CW. Comparative metabolism of codeine in man, rat, dog, guinea-pig and rabbit: identification of four new metabolites. J Pharm Pharmacol. 1979 May;31(5):314-7. doi: 10.1111/j.2042-7158.1979.tb13507.x. PMID 37301
- [Background] Otton SV, Schadel M, Cheung SW, Kaplan HL, Busto UE, Sellers EM. CYP2D6 phenotype determines the metabolic conversion of hydrocodone to hydromorphone. Clin Pharmacol Ther. 1993 Nov;54(5):463-72. doi: 10.1038/clpt.1993.177. PMID 7693389

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Group 1 | Group 2
Started | 16 | 14
Completed | 15 | 14
Not Completed | 1 | 0
Not completed — Physician Decision | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 | Group 2 | Total
Number analyzed (Participants) | 16 | 14 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.63 (8.937) | 54.28 (8.279) | 48.60 (10.062)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 10 | 21
  Male | 5 | 4 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 16 | 13 | 29
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 15 | 13 | 28
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 16 | 14 | 30

OUTCOME MEASURES:

1. Primary Outcome: Peak Plasma Concentration of Hydromorphone
Description: Determine the plasma pharmacokinetic profile of hydromorphone in chronic pain subjects taking hydrocodone within a 6 hour time frame. Note: Sensitivity of the lab test used to determine plasma hydromorphone concentrations was not sufficient. Failure to meet the lowest level of detection, all subjects plasma hydromorphone concentrations were recorded as zero at all time points.
Time Frame: Up to 6 hours
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 16 | 14
ng/mL
  Hour 0 | 0 (0) | 0 (0)
  Hour 1 | 0 (0) | NA (NA) — No blood drawn at this time point
  Hour 2 | NA (NA) — No blood drawn at this time point | 0 (0)
  Hour 3 | 0 (0) | NA (NA) — No blood drawn at this time point
  Hour 4 | NA (NA) — No blood drawn at this time point | 0 (0)
  Hour 5 | 0 (0) | NA (NA) — No blood drawn at this time point
  Hour 6 | NA (NA) — No blood drawn at this time point | 0 (0)

2. Secondary Outcome: Correlation of Plasma PK of Hydrocodone
Description: Correlate the plasma pharmacokinetic profile of hydromorphone to their hydrocodone doses.
Time Frame: 1 Month
Population: Analysis could not be performed because plasma levels analyzed were too low for the assay chosen.
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Peak Urine Concentration of Hydromorphone
Description: Analyze the urine concentration of hydromorphone
Time Frame: Up to 4 hours
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 16 | 14
ng/mL
  Hour 0 | 726.69 (1294.77) | 211.36 (248.356)
  Hour 3 | 815.63 (1396.38) | NA (NA) — No urine was taken at this time point.
  Hour 4 | NA (NA) — No urine was taken at this time point. | 205.57 (239.508)

ADVERSE EVENTS:
Time Frame: From time of first dose of Hydrocodone to Completion of study.
Arm/Group | Group 1 | Group 2
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/14
Other Adverse Events (participants affected / at risk) | 0/16 | 0/14

LIMITATIONS AND CAVEATS:
Sensitivity of the lab test used to determine plasma hydromorphone concentrations was not sufficient. Failure to meet the lowest level of detection, all subjects plasma hydromorphone concentrations were recorded as zero at all time points.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No